CLINICAL TRIAL: NCT00600613
Title: A Pilot Study to Assess the Feasibility of Cone Beam CT to Localize Liver Metastases Immediately Prior to Radiotherapy
Brief Title: Assess the Feasibility of Cone Beam CT to Localize Liver Metastases Immediately Prior to Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 05-129
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Results first posted 2015-04-17 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-04

CONDITIONS: Localize Liver Metastases
Keywords: Radiation Therapy

ARMS (1):
- 1 (Experimental): Patients going for treatment of liver metastases with radiation therapy.
  Interventions: Radiation: cone beam imaging

INTERVENTIONS:
Radiation: cone beam imaging — All study patients will undergo simulation, treatment planning and verification as currently practiced. The contrast injection and cone beam imaging will be added to the standard procedure just prior to treatment delivery on the first and last days of treatment only.

SUMMARY:
The purpose of this study is to test a new and possibly more accurate method of positioning patients with liver tumors in preparation for radiation treatment.

The positioning of patients with liver cancer is important because the tumor moves a bit when you breathe and makes it hard to determine the right position of the tumor at the time of treatment. Also, depending upon what is in your stomach at the time of treatment, it may change the shape of the liver and make it difficult to plan the radiation treatment. As part of this study, we will take a new type of image of your liver in addition to the standard portal images. This new type of image is called a cone-beam image. It shows a much more detailed picture of the liver tumors than the standard portal images. Normally, marker seeds need to be placed near the liver metastasis for radiation treatment. If the results of this study show that the tumor can be positioned as accurately with the new images as with the old images, then future patients with liver tumors would not have to have marker seeds placed into their liver. The use of cone beam imaging for the setup of patients with liver tumors is new.

ELIGIBILITY:
Inclusion Criteria:

* Age > than or equal to 18 years
* KPS > than or equal to 80
* Able to tolerate immobilization cradle positioning
* Able to give informed consent
* Histologically confirmed diagnosis of solid tumor malignancy
* Liver metastases visualized on CT imaging

Exclusion Criteria:

* Lymphoid primary histology (lymphoma/leukemia)
* Allergic reaction to intravenous CT contrast
* Liver function tests (AST, ALT, Bilirubin) > 2.0 x normal
* Abnormal kidney function (serum creatinine > 1.5)
* INR > 2.0, Platelet count <70.000.
* Marker seed placement not possible
* > 5mm excursion after abdominal compression

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiya Yamada, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Going for Treatment of Liver Metastases With RT: Patients going for treatment of liver metastases with radiation therapy.
Period: Overall Study
Arm/Group | Patients Going for Treatment of Liver Metastases With RT
Started | 6
Completed | 5
Not Completed | 1
Not completed — Protocol Deviation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients Going for Treatment of Liver Metastases With RT
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Eligible for Cone Beam Tumor Localization"
Description: Assess the feasibility of using a new imaging technique called "cone beam imaging" to localize a liver tumor immediately prior to external beam radiotherapy.
Time Frame: Up to 2 hours
Measure: Number; unit: participants
Arm/Group | Patients Going for Treatment of Liver Metastases With RT
Number analyzed (Participants) | 5
participants | 5

ADVERSE EVENTS:
Arm/Group | Patients Going for Treatment of Liver Metastases With RT
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes